CLINICAL TRIAL: NCT06906666
Title: Analysis of Injury Risk Factors in Elite Athletes. A Cross-sectional Cohort Study.
Brief Title: Analysis of Injury Risk Factors in Elite Athletes
Status: Completed | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Ruben Cuesta Barriuso, Principal Investigator, University of Oviedo
Other Study IDs: ATL-risk
Record Dates: First submitted 2025-03-25; First posted 2025-04-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-03

CONDITIONS: Athletic Injuries
Keywords: Muscle Injury; Athletics; Risk; Secondary Prevention; Physiotherapy
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observacional group
  Interventions: Other: Athletes sample

INTERVENTIONS:
Other: Athletes sample — Elite athletes in whom the risk of injury will be calculated and the influence of confounding factors will be assessed through a personal interview.
  Other Names: Elite athletes group

SUMMARY:
Background information. The different disciplines of athletics place high physical demands on athletes. These different categories of running vary in terms of physical effort and duration, generating different levels of risk of injury. The description of the main injuries that affect elite athletes in the different athletics disciplines, as well as the identification of the specific risk factors of each discipline, will allow the identification of preventive measures to be implemented.

Objective. To identify the risk factors for tendon injury in professional long- and middle-distance athletes, according to the type of event, and to identify the best predictive model for tendon injuries based on anthropometric and athletic variables.

Method. Ambispective cohort study. 81 elite athletes will be recruited. The primary variable will be the number of tendon injuries in the last three seasons. The secondary and modifying variables will be: age (in completed years), weekly training load (in minutes), type of footwear (sneakers without carbon plate, sneakers with carbon plate, spiked sneakers without carbon plate and spiked sneakers with carbon plate), diet (balanced, high in carbohydrates, high-protein, controlled hypocaloric and adapted to the training cycle) and the regular practice of another physical activity. The possible confounding variables will be the body mass index, the date of tendon injuries in that period and the time spent as a federated athlete (in completed months). The analysis will calculate the risk of injury in these athletes and assess the influence of confounding factors and trend analysis on the primary variable, stratified by possible confounding factors.

Expected results. To calculate the risk of injury in elite athletes based on anthropometric and sociodemographic variables. To identify the predictive model of tendon injuries in elite athletes

ELIGIBILITY:
Inclusion Criteria:

* Elite federated athletes
* Who have not undergone previous musculoskeletal surgery in the seasons under study
* Who were federated at least one year before the study period
* Sign the informed consent document.

Exclusion Criteria:

* Athletes who have not participated in competition, during the study seasons, for a period of more than 6 months due to a musculoskeletal injury

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Elite athletes
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Measurement of number of lower limb tendon injuries | Screening visit
  The primary variable will be the number of lower limb tendon injuries in the last three seasons

SECONDARY OUTCOMES:
Measurement of age | Screening visit
  The measurement of age (measured in completed years) will be a secondary variable.
Measurement of the weekly training load | Screening visit
  The measurement of the weekly training load (measured in minutes) will be a secondary variable.
Measurement of the type of footwear | Screening visit
  The evaluation of the type of footwear (with the response options: shoe without carbon plate, shoe with carbon plate, spike shoe without carbon plate and spike shoe with carbon plate) will be a secondary variable.
Measurement of the type of diet | Screening visit
  The evaluation of the type of diet (with the response options: balanced, rich in carbohydrates, rich in proteins and adapted to the training cycle) will be a secondary variable.
Measurement of the practice of another physical activity | Screening visit
  The evaluation of the practice of another physical activity on a regular basis will be a secondary variable.

OTHER OUTCOMES:
Measurement of the body mass index | Screening visit
  The measurement of the body mass index (measured in kg/m2) will be a possible confounding variable.
Measurement of the date of tendon injuries | Screening visit
  The date of tendon injuries in that period will be a possible confounding variable.
Measurement of federated time | Screening visit
  The evaluation of federated time (measured in completed months) will be a possible confounding variable.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, Study Director — Universidad de Oviedo
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: Undecided